CLINICAL TRIAL: NCT04879368
Title: A Randomised Phase III Open Label Study of Regorafenib + Nivolumab vs Standard Chemotherapy in Refractory Advanced Gastro-Oesophageal Cancer (AGOC)
Brief Title: RegoNivo vs Standard of Care Chemotherapy in AGOC
Acronym: INTEGRATEIIb
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: Bayer (Industry); Bristol-Myers Squibb (Industry); University of Sydney (Other); Academic and Community Cancer Research United (Other); Taiwanese Cooperative Oncology Group (Unknown); Frankfurter Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Unknown); National Cancer Center Hospital East (Other); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0315OG/CTC0140; 2020-004617-12 (EudraCT Number)
Record Dates: First submitted 2021-02-24; First posted 2021-05-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Gastro-Oesophageal Cancer
Keywords: Metastatic; Locally recurrent; Oesophago-gastric junction; Stomach; Adenocarcinoma; Undifferentiated carcinoma; RegoNivo
MeSH Terms: conditions — Neoplasm Metastasis; Adenocarcinoma; Carcinoma | interventions — regorafenib; Nivolumab; Docetaxel; Paclitaxel; Albumin-Bound Paclitaxel; Irinotecan; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RegoNivo (Experimental): Participants in the RegoNivo arm will;
  1. self-administer 90mg (3x30mg) of regorafenib days 1-21 of each 28-day treatment cycle and;
  2. receive intravenous nivolumab 240 mg day 1 of each 14 day cycle until disease progression or prohibitive adverse events as per protocol, given in hospital by infusion.
  After 2 months, patients whose disease is controlled may have nivolumab administered 480 mg every 28 days.
  Interventions: Drug: Regorafenib; Biological: Nivolumab
- Standard of Care (Active Comparator): Participants in the control arm will receive investigator choice chemotherapy with any of the following agents
  * taxane (paclitaxel or docetaxel)
  * irinotecan or
  * oral trifluridine/tipiracil (TAS102)
  All treatment groups will receive Best Supportive Care (BSC).
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Irinotecan; Drug: Trifluridine/Tipracil

INTERVENTIONS:
Drug: Regorafenib — Oral multi-targeted tyrosine kinase inhibitor (TKI) which targets angiogenic (VEGF, TIE-2), stromal (PDGF-β), and oncogenic (RAF, RET and KIT) receptor tyrosine kinases
  Other Names: Stivarga
  Arms: RegoNivo
Biological: Nivolumab — human IgG4 monoclonal antibody inhibitor of PD-1
  Other Names: Opdivo
  Arms: RegoNivo
Drug: Docetaxel — Docetaxel is taxane-derivative chemotherapy drug, used in the treatment of early, locally advanced and metastatic breast cancer. It is an anti-microtubule agent. Other uses are in the treatment of non-small cell lung cancer, advanced stomach cancer, head and neck cancers, soft tissue sarcoma, ovarian cancer, metastatic prostate cancer, etc.
  microtubules, and simultaneously promotes assembly and inhibits disassembly of them
  Other Names: Taxotere
  Arms: Standard of Care
Drug: Paclitaxel — Paclitaxel is one of several cytoskeletal drugs that target tubulin. Paclitaxel-treated cells have defects in mitotic spindle assembly, chromosome segregation, and cell division. Unlike other tubulin-targeting drugs, such as colchicine, that inhibit microtubule assembly, paclitaxel stabilizes the microtubule polymer and protects it from disassembly. Chromosomes are thus unable to achieve a metaphase spindle configuration. This blocks the progression of mitosis and prolonged activation of the mitotic checkpoint triggers apoptosis or reversion to the G0-phase of the cell cycle without cell division
  Other Names: Abraxane
  Arms: Standard of Care
Drug: Irinotecan — Camptothecin, one of the four major structural classifications of plant-derived anti-cancerous compounds, is a cytotoxic alkaloid which consists of a pentacyclic ring structure containing a pyrrole (3, 4 β) quinoline moiety, an S-configured lactone form, and a carboxylate form. Irinotecan is activated by hydrolysis to SN-38, an inhibitor of topoisomerase I. This is then inactivated by glucuronidation by uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1). The inhibition of topoisomerase I by the active metabolite SN-38 eventually leads to inhibition of both DNA replication and transcription.
  Other Names: Camptosar
  Arms: Standard of Care
Drug: Trifluridine/Tipracil — The drug consists of the cytotoxin trifluridine and the thymidine phosphorylase inhibitor (TPI) tipiracil. Trifluridine is incorporated into DNA during DNA synthesis and inhibits tumor cell growth. Trifluridine (TFT) is incorporated into DNA by phosphorylation by thymidylate kinase (TK) to TF-TMP; TF-TMP then covalently binds to tyrosine 146 of the active site of thymidylate synthase (TS) inhibiting the enzyme's activity. TS is vital to the synthesis of DNA because it is an enzyme involved in the synthesis of the deoxynucleotide, thymidine triphosphate (dTTP). Inhibition of TS depletes the cell of dTTP and causes accumulation of deoxyuridine monophosphate (dUMP), which increases the likelihood that uracil gets misincorporated into the DNA.
  Other Names: Lonsurf
  Arms: Standard of Care

SUMMARY:
To determine if the regorafenib and nivolumab combination (RegoNivo) improves overall survival compared with current standard chemotherapy options in refractory AGOC.

DETAILED DESCRIPTION:
The purpose of this international study is to determine if the combination of regorafenib and nivolumab is more effective than standard chemotherapy in prolonging overall survival in a broad group of participants with AGOC, who have progressed after treatment with standard anti-cancer therapy.

In the INTEGRATE study, regorafenib alone was shown to be effective in prolonging the progression-free period in people with AGOC following standard anti-cancer therapy (i.e. it delayed tumour growth), and demonstrated a potential benefit on long term survival. Recent research has shown the early results from this combination of regorafenib & nivolumab may improve outcomes for cancer patients. INTEGRATE IIb will investigate this effect further in a larger group of participants with AGOC.

The study aims to determine:

i. Whether the combination of regorafenib/nivolumab is likely to help patients with AGOC live longer; ii. The effects of this treatment on progression-free survival; iii. The numbers of participants responding to the treatment iv. The effects of this treatment on quality of life v. The side effects and tolerability of this treatment vi. Molecular differences (e.g. variations in genes or proteins) that may account for the effects of this treatment vii. Differences in the costs of care for people on this treatment.

The Investigators plan to enrol 460 participants in the study from, but not limited to; Australia, South Korea, Japan, Taiwan, USA, Germany, Austria, Spain, and Italy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years or over) with metastatic or locally recurrent gastro-oesophageal cancer which:

   1. has arisen in any primary gastro-oesophageal site (oesophago-gastric junction (GOJ) or stomach); and
   2. is of adenocarcinoma or undifferentiated carcinoma histology; and
   3. is evaluable according to Response Evaluation Criteria in Solid Tumours (RECIST Version 1.1) by computed tomography (CT) scan performed within 21 days prior to randomisation. A lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of the lesion prior to study enrolment; and
   4. has failed or been intolerant to a minimum of 2 lines of prior anti-cancer therapy for recurrent/metastatic disease which must have included at least one platinum agent and one fluoropyrimidine analogue. Note: Neoadjuvant or adjuvant chemotherapy or chemoradiotherapy will be considered as first line treatment where people have relapsed or progressed within 6 months of completing treatment; Radiosensitising chemotherapy given solely for this purpose concurrent with palliative radiation will not be considered as a line of treatment. Ramucirumab monotherapy, or immunotherapy with a checkpoint inhibitor, will be considered a line of treatment.
   5. HER2-positive participants must have received trastuzumab
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (Appendix 1).
3. Ability to swallow oral medication.
4. Adequate bone marrow function (Platelets ≥100x109/L; Absolute Neutrophil Count (ANC) ≥1.5x109/L and Haemoglobin ≥ 9.0g/dL).
5. Adequate renal function (Creatinine clearance >50 ml/min) based on either the Cockcroft-Gault formula (Appendix 2), 24-hour urine or Glomerular Filtration Rate (GFR) scan; and serum creatinine ≤1.5 x Upper Limit of Normal (ULN).
6. Adequate liver function (Serum total bilirubin ≤1.5 x ULN, and INR ≤ 1.5 x ULN, and Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP) ≤2.5 x ULN (≤ 5 x ULN for participants with liver metastases)).

   Participants being treated with an anti-coagulant, such as warfarin or heparin, will be allowed to participate provided that no prior evidence of an underlying abnormality in these parameters exists.
7. Willing and able to comply with all study requirements, including treatment, timing, and/or nature of required assessments and follow-up.
8. Study treatment both planned and able to start within 7 days after randomisation (note: subjects randomised on a Friday should commence treatment no earlier than the following Monday)
9. Signed, written informed consent

Exclusion Criteria:

1. Known allergy to the investigational product drug class or excipients in the regorafenib and/or nivolumab
2. Poorly-controlled hypertension (systolic blood pressure >140mmHg or diastolic pressure> 90mmHg despite optimal medical management).
3. Participants with known, uncontrolled malabsorption syndromes
4. Any prior anti-VEGF targeted therapy using small molecule VEGF TKIs (e.g. apatinib). Prior anti-VEGF targeted monoclonal antibody therapies (e.g. bevacizumab and ramucirumab) are permitted.
5. Any prior use of more than one immune checkpoint inhibitor
6. Treatment with any previous drug therapy within 2 weeks prior to first dose of study treatment. This includes any investigational therapy.
7. Use of biological response modifiers, such as granulocyte colony stimulating factor (G-CSF), within 3 weeks prior to randomisation.
8. Concurrent treatment with strong CYP3A4 inhibitors or inducers.
9. Palliative radiotherapy, unless more than 14 days have elapsed between completion of radiation and the date of registration, and adverse events resulting from radiation have resolved to < Grade 2 according to CTCAE V5.0
10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization
11. Arterial thrombotic or ischaemic events, such as cerebrovascular accident, within 6 months prior to randomization.
12. Venous thrombotic events and pulmonary embolism within 3 months prior to randomization
13. Any haemorrhage or bleeding event ≥ Grade 3 according to CTCAE v5.0 within 4 weeks prior to randomization.
14. Non-healing wound, ulcer, or bone fracture.
15. Interstitial lung disease with ongoing signs and symptoms
16. Clinical hyperthyroidism or hypothyroidism. Note: non-clinically significant abnormal TFTs (abnormal TSH and abnormal T3 and/or abnormal T4) considered to be due to sick euthyroid syndrome is allowed.
17. Persistent proteinuria of ≥ Grade 3 according to CTCAE v5.0 (equivalent to > 3.5g of protein over 24 hour measured on either a random specimen or 24 hour collection.
18. Uncontrolled metastatic disease to the central nervous system. To be eligible, known CNS metastases should have been treated with surgery and/or radiotherapy and the patient should have been receiving a stable dose of steroids for at least 2 weeks prior to randomization, with no deterioration in neurological symptoms during this time.
19. History of another malignancy within 2 years prior to randomization. Participants with the following are eligible for this study:

    1. curatively treated cervical carcinoma in situ,
    2. non-melanomatous carcinoma of the skin,
    3. superficial bladder tumours (T1a [Non-invasive tumour], and Tis [Carcinoma in situ]),
    4. treated thyroid papillary cancer
20. Any significant active infection, including chronic active hepatitis B, hepatitis C, or HIV. Testing for these is not mandatory unless clinically indicated. Participants with known Hepatitis B/C infection will be allowed to participate providing evidence of viral suppression has been documented and the patient remains on appropriate anti-viral therapy.
21. Patients with acute coronary syndrome (including myocardial infarction and unstable angina), and with a history of coronary angioplasty or stent placement performed within 6 months before enrolment
22. Patients with a ≥ grade 3 active infection according to CTCAE version 5.0
23. Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease
24. Patients who require systemic corticosteroids (excluding temporary usage for tests, prophylactic administration for allergic reactions, or to alleviate swelling associated with radiotherapy; if used as replacement therapy e.g. ≤ 10 mg prednisolone or dexamethasone ≤ 2 mg per day) or immunosuppressants, or who have received such a therapy < 14 days prior to randomisation
25. Patients with a seizure disorder who require pharmacotherapy
26. Serious medical or psychiatric condition(s) that might limit the ability of the patient to comply with the protocol.
27. Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to randomization. Men must have been surgically sterilized or use a barrier method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
O/S | 5 years
  To determine the effect of RegoNivo on overall survival (OS) (death from any cause) in the overall study population and in the Asian sub-population.

SECONDARY OUTCOMES:
Determine the effect of RegoNivo on; PFS | 5 years
  Progression free survival (PFS)(disease progression or death) in the study population
Determine the effect of RegoNivo on; OTRR | 5 years
  Objective tumour response rate (OTRR)((partial or complete response (PR or CR)) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and iRECIST on study population
Determine the effect of RegoNivo on; QoL - EORTC Quality of Life Questionnaire | 5 years
  Quality of life (QoL)(scores from participant-completed questionnaires) of participants on study EORTC QLQ-C30: Q1 - Q28, Min 1 Max 4, Higher Score = Worse
Determine the effect of RegoNivo on; QoL - EORTC Quality of Life Questionnaire | 5 years
  Quality of life (QoL)(scores from participant-completed questionnaires) of participants on study EORTC QLQ-C30: Q29 & Q30 Min 1 Max 7, Higher = Better
Determine the effect of RegoNivo on; QoL - EORTC Quality of Life Questionnaire -Stomach Cancer | 5 years
  Quality of life (QoL)(scores from participant-completed questionnaires) of participants on study EORTC QLQ STO22 Min 1 Max 4, Higher Score = Worse
Determine the effect of RegoNivo on; QoL - Patient D.A.T.A form (self assessment of pain on health aspect) | 5 years
  Quality of life (QoL)(scores from participant-completed questionnaires) of participants on study Patient D.A.T.A Form: Q1 - Q17 Min 0 Max 10, Higher Score = Worse
Determine the effect of RegoNivo on; QoL - Patient D.A.T.A form (self rating on health aspects) | 5 years
  Quality of life (QoL)(scores from participant-completed questionnaires) of participants on study Patient D.A.T.A Form: Q18 - Q24 Min 0 Max 10, Higher Score = Better
Determine the effect of RegoNivo on; QoL - Patient D.A.T.A form (health aspect impact self assessment) | 5 years
  Quality of life (QoL)(scores from participant-completed questionnaires) of participants on study Patient D.A.T.A Form: Q25 - Q47 Min 0 Max 10, Higher Score = Worse
Determine the effect of RegoNivo on; QoL - Health Questionnaire | 5 years
  Quality of life (QoL)(scores from participant-completed questionnaires) of participants on study EQ-5D-5L Health questionnaire Min 0 Max 100, Higher Score = Better
Determine the effect of RegoNivo on; Safety | 5 years
  Safety (rates of adverse events) of participants on study

OTHER OUTCOMES:
Prognostic biomarker identification for AGOC | Up to 24 months following close of study.
  To identify prognostic and predictive biomarkers (tissue and circulating) for study endpoints (relating to survival, response and safety).
Regorafenib max plasma concentration level assessment (Cmax) across geographical regions | Up to 24 months following close of study.
  To evaluate regorafenib Cmax in patient populations from different geographical regions (regorafenib levels).
Regorafenib levels and correlation to treatment | Up to 24 months following close of study.
  To evaluate regorafenib levels and their correlation to outcomes in treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nick Pavlakis, Prof, Study Chair — AGITG
Locations (94):
- United States (6):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - USC Norris, Los Angeles, California
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - St Elizabeth Healthcare, Edgewood, Kentucky
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Fred Hutchinson Cancer Research Centre - South Lake Union Clinic, Seattle, Washington
- Australia (24):
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St Vincent's Public Hospital, Darlinghurst, New South Wales
  - Border Medical Oncology Research Unit, East Albury, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Private Hospital, Sydney, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Ballarat Oncology and Haematology Services, Wendouree, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - The Townsville Hospital, Douglas, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Sunshine Coast University Hospital, Sunshine Coast, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health, Clayton, Victoria
  - Austin Health, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St John of God Hospital Subiaco, Subiaco, Western Australia
- Austria (4):
  - Landeskrankenanstalten-Betriebsgesellschaft-KABEG, Klagenfurt
  - Ordensklinikum Linz GmbH Barmherzige schwestern, Linz
  - Medizinische Universitaet Wien, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Germany (22):
  - Evang. Klinikum Bethel Bielefeld, Gütersloh, North Rhine-Westphalia
  - Helios Bad Saarow, Bad Saarow
  - Klinikum Bayreuth, Bayreuth
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Kliniken der Stadt Köln, Cologne
  - KEM/Evang. Kliniken Essen Mitte gGmbH, Essen
  - Institut für Klinisch Onkol Forschung am Krankenhaus Nordwest, Frankfurt
  - Universitätsklinikum Greifswald, Greifswald
  - Norddeutsches Studienzentrum für Innovative Onkologie (NIO), Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Klinikum Ludwigburg, Ludwigsburg
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Universitätsklinikum Mainz, Mainz
  - Philipps-Universitat Marburg, Marburg
  - Klinikum rechts der Isar der TU München, München
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Caritas Klinikum Saarbrücken St. Theresia, Saarbrücken
  - Universitätsklinikum Ulm, Ulm
- Italy (6):
  - Istituto Nazionale Tumori di Napoli-IRCCS Fondazione G. Pascale, Napoli
  - Universitae degli studi della Campania "Luigi Vanvitelli", Napoli
  - Azienda USL-IRCCS Di Reggio Emilia, Reggio Emilia
  - San Camillo Forlanini Hospitals, Roma
  - Universita Cattolica del Sacro Cuore, University Hospital Gemelli, Roma
  - IRCCS Fondazione Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Japan (6):
  - National Cancer Centre Hospital East, Chiba, Kashiwa
  - Hokkaido University Hospital, Sapporo, Kita
  - Kyushu Cancer Center, Fukuoka
  - Shikoku Cancer Center, Matsuyama
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
- South Korea (18):
  - Hallym University Sacred Heart Hospital, Anyang
  - Dong-A University Hospital, Busan
  - Haeundae Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Asan Medical Centre, Seoul
  - Chung-Ang University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea - Yeouido St. Mary's Hospital, Seoul
  - Yonsei University Health System - Gangnam Severance Hospital, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Clinico Universitario De Valencia, Valencia
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital (CMUH), Taichung
  - National Cheng Kung University Hospital, Taipei
  - National Taiwan University Hospital (NTUH), Taipei
  - Taipei Veterans General Hospital (TPVGH), Taipei

REFERENCES:
- [Derived] Lam LL, Pavlakis N, Shitara K, Sjoquist KM, Martin AJ, Yip S, Kang YK, Bang YJ, Chen LT, Moehler M, Bekaii-Saab T, Alcindor T, O'Callaghan CJ, Tebbutt NC, Hague W, Chan H, Rha SY, Lee KW, Gebski V, Jaworski A, Zalcberg J, Price T, Simes J, Goldstein D. INTEGRATE II: randomised phase III controlled trials of regorafenib containing regimens versus standard of care in refractory Advanced Gastro-Oesophageal Cancer (AGOC): a study by the Australasian Gastro-Intestinal Trials Group (AGITG). BMC Cancer. 2023 Feb 22;23(1):180. doi: 10.1186/s12885-023-10642-7. PMID 36814222